CLINICAL TRIAL: NCT04810728
Title: Efficacy of Psidii Guava's Extract For Mild And Symptomless Coronavirus Disease-19 (COVID-19)
Brief Title: Efficacy of Psidii Guava's Extract For COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Faculty of Medicine Baiturrahmah University (Other)
Responsible Party: Principal Investigator, Fredia Heppy, MD, SpPD, FINASIM, Lecturer of Internal Medicine, Prinsipal Investigator, Faculty of Medicine Baiturrahmah University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSIDII0520_COV19
Record Dates: First submitted 2021-03-16; First posted 2021-03-23 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Covid19
Keywords: Psidii guava extract; Coronavirus Disease-19
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extract Psidii guava (Experimental): 2 Capsule of extract Psidii guava, three times daily
  Interventions: Drug: Extract Psidii guava; Combination Product: Standard therapy for Covid-19 patient
- Standard therapy (Active Comparator): Standard therapy for Covid-19 patient (vitamin C, Zinc, medication for clinical symptoms such as: antipyretic agent, decongestan and mucolytic.)
  Interventions: Combination Product: Standard therapy for Covid-19 patient

INTERVENTIONS:
Drug: Extract Psidii guava — 2 Capsule Extract Psidii guava, three times daily
  Other Names: Psidii
  Arms: Extract Psidii guava
Combination Product: Standard therapy for Covid-19 patient — (Vitamin C, Zinc, medication for clinical symptoms such as: antipyretic agent, decongestan and mucolytic.)

SUMMARY:
This study was an experimental, randomized clinical trial, with a parallel design, with aims were seeing the effectiveness of extracted Psidii guava on white blood cells (WBCs) count, neutrophil, lymphocyte, monocyte, neutrophil-lymphocyte ratio (NLR), high sensitive C reactive protein (hs-CRP), proportion and duration COVID-19 seroconversion subjects compared to controls.

One of the herbs standardized that was commonly used in Indonesia is extracted Psidii guava, which is known as a guava leaf extract. Extract Psidii guava contains chemical substances saponins, oleanolic acid, xylopyranoside, flavonoids, quercetin, arabinopyranoside, and Guaijavarin. The Previous study on Psidii guava stated that guava leaves contain lots of flavonoids, especially quercetin. An in vitro study of dengue virus type 2 found that quercetin significantly inhibited the activity of the DEN-2 virus, while other flavonoids looked weaker. On the other hand, in an in vitro test of glycosylated flavonoids from Psidium Geunesse, which is a guava leaf from Brazil, received the use of flavonoids in Psidium Geunesse to inhibit HIV-1 virus activity with a 50% inhibition concentration of about 8.5 μg / ml compared to single active substances. Quercetin with a 50% inhibitory concentration of about 53μg / ml. These flavonoids also inhibited the enzyme reverse transcriptase HIV-1(RT)with an inhibition concentration of 7.2 μM compared to quercetin 0.6 μM single. Another study found that quercetin in Psidii guava inhibits RNA polymerase, which is important in dengue virus replication. In addition, quercetin can inhibit protease enzyme, helicase domain, and viral ATPase enzyme.

There is an antiviral effect based on limited in vitro studies but with quite a lot of literature studies, and considering that there are no effective antiviral drugs against COVID-19, especially mild and moderate cases, also considering the length of healing time for patients COVID-19 with the risk of isolation. For a long time with various consequences, researchers tried to examine the effectiveness of extract Psidii guava inpatients COVID-19 at the quarantine location of the West Sumatra Provincial Government. Extract Psidii guava is hypothesized to improve WBCs, neutrophil, lymphocyte, monocyte, NLR, hs-CRP level, to increase proportion and shorten the duration of COVID-19 seroconversion in mild and symptomless cases.

DETAILED DESCRIPTION:
There will be 2 groups of treatment; each group will consist of 45 subjects with the treatment regimens maximal for 4 weeks.

The treatment I: 2 capsules of Extract Psidii guava, three times daily. Treatment II: standard therapy for Covid-19 patient (vitamin C, Zink, medication for clinical symptoms such as antipyretic agent, decongestant, and mucolytic).

The eligible subjects will be randomly allocated to receive study medication (Treatment 1 or Treatment 2) for 7 days, if the result swab after treatment still positive, patients will be given extract Psidii guava capsule with the same dose till maximal 4 weeks. Treatment Group 1 will receive 2 capsules of Extract Psidii guava, three times daily. While Treatment Group 2 will receive the standard therapy for Covid-19 patient.

Subjects will be evaluated for treatment efficacy at baseline 7 days after treatment and 28 days (4 weeks) treatment. The demographic profile, such as age and sex, will be measured at baseline. White blood cells count, neutrophil, lymphocyte, monocyte, NLR, hs-CRP level at baseline and 7 days after treatment, while proportion and duration COVID-19 seroconversion will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Confirmed positive COVID-19 mild and symptomless
* Aged 13 - 59 years
* Willing to take part in the study and sign an informed consent

Exclusion Criteria:

* Not willing to join the study
* History of allergy to the research drug (extract Psidii guava)

Ages: 13 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Changes of inflammatory cells and marker | 7 days (1 week)
  1. Leucocyte count in mm3
  2. Neutrophil count in %
  3. Lymphocyte count in %
  4. Monocyte count in %
  5. Neutrophil-lymphocyte ratio
  6. High sensitivity C reactive protein in ng/mL

SECONDARY OUTCOMES:
Recovery rate | 14 days (2 weeks), maximal 28 days (4 weeks)
  Recovery proportion patients with COVID-19 mild and symptompless cases at the end of study
Duration of seroconversion | Maximal 28 days
  Length of conversion detected of RT PCR RNA virus of SARS-COV-19 from positive to negative

CONTACTS AND LOCATIONS:
Overall Officials: Fredia Heppy, MD, FINASIM, Principal Investigator — Faculty of Medicine, Baiturrahmah University, Padang, West Sumatera, Indonesia
Locations (1):
- Faculty of Medicine, Baiturrahmah University, Padang, West Sumatera, Indonesia

REFERENCES:
- [Derived] Heppy F, Mulyana R, Afrainin Syah N, Tjandrawinata RR. The effect of Psidium guajava Leaves' extract for mild and asymptomatic corona virus Disease-19. Saudi Pharm J. 2023 Apr;31(4):592-596. doi: 10.1016/j.jsps.2023.02.012. Epub 2023 Mar 7. PMID 37009425